CLINICAL TRIAL: NCT03047551
Title: Is Transabdominal Sonography Comparable to Transvaginal Sonography for Eligibility Assessment Prior to Medical Abortion? A Randomized Controlled Trial.
Brief Title: Transabdominal and Transvaginal Sonography in Medical Abortion
Acronym: TASvTVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Carolyn Westhoff, Professor of Obstetrics and Gynecology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAQ8722
Record Dates: First submitted 2016-10-24; First posted 2017-02-09 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Abortion Early
Keywords: Abortion, induced; Ultrasonography; Health Services accessibility; Pragmatic Clinical Trial; Randomized controlled trial as topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transabdominal Sonography (Active Comparator): Subjects will receive transabdominal sonography using a standard ultrasound device to determine medical abortion eligibility.
  A transabdominal ultrasound is used to look at the pelvic organs. Gel is placed on your abdomen. Then a small, handheld unit called a transducer is gently moved around to view the pelvic organs. The transducer sound waves make a picture on the TV screen.
  Interventions: Procedure: Transabdominal sonography
- Transvaginal Sonography (Active Comparator): Subjects will receive transvaginal sonography using a standard ultrasound device to determine medical abortion eligibility.
  Transvaginal ultrasound is an examination of the female pelvis and urogenital tract (kidneys and bladder). It differs from an abdominal ultrasound as it looks at the pelvic organs from inside the vagina.
  Interventions: Procedure: Transvaginal sonography

INTERVENTIONS:
Procedure: Transabdominal sonography — Ultrasound machines vary by site. At Planned Parenthood and Columbia University Medical Center, providers utilize the LOGIQ P5 ultrasound machine, manufactured by General Electric Healthcare.
  Other Names: TAS
  Arms: Transabdominal Sonography
Procedure: Transvaginal sonography — Ultrasound machines vary by site. At Planned Parenthood and Columbia University Medical Center, providers utilize the LOGIQ P5 ultrasound machine, manufactured by General Electric Healthcare.
  Other Names: TVS
  Arms: Transvaginal Sonography

SUMMARY:
The investigator will perform a multicenter, randomized controlled trial in practices that routinely use transvaginal sonography (TVS) to compare how often clinicians order additional testing prior to medical abortion after the use of either TVS or transabdominal ultrasound (TAS) in medical abortion eligibility assessment. Women will be randomized to receive either TVS or TAS prior to medical abortion. We anticipate enrolling 800 patients receiving care from about 30 providers over 6-8 months.

The primary study outcome will be the proportion of women that requires additional evaluation after sonography, prior to determination of medical abortion eligibility. The second primary outcome will be patient satisfaction, determined by a patient satisfaction questionnaire utilizing a visual analog scale.

DETAILED DESCRIPTION:
Ultrasound use in the assessment of medical abortion eligibility varies by practice site. The National Abortion Federation (NAF), the Society of Family Planning (SFP), and the World Health Organization (WHO) guidelines do not recommend routine use of sonography; however, many institutions and practices still require this as part of clinic protocol. Many clinicians routinely perform transvaginal sonography (TVS), a more invasive assessment than transabdominal ultrasound (TAS); reliance on TVS, specifically, can be cost-prohibitive due to high-level disinfection (HLD) requirements. Thus, routine US use can greatly decrease access to abortion services.

Medical abortion accounts for an increasing proportion of abortions performed in the United States; as of 2012, 20.8% of all abortions were medical abortions. Routine use of ultrasonography and particularly TVS may be a holdover secondary to its use in early clinical trials of medical abortion efficacy - its use has remained a part of many providers' clinical practice despite evidence that it is not always necessary.

This study, specifically, would be of value for the many clinicians who currently use TVS for all medical abortion patients and could support using TAS rather than TVS in a majority of these patients. The results could also provide guidance on how often practice settings without TVS and HLD would be able to provide medical abortion, and for which patients. Such settings could include primary care or rural clinics, any low volume clinics, or those where the costs and time associated with the HLD required for use of TVS prohibit or limit the provision of medical abortion. In addition, even high-volume specialty family planning clinics would benefit from a reduction in use of TVS. In the US, many providers have sonography available and use it routinely. However, even in the US, many clinics may seek to offer medical abortion without sonography, and other researchers are studying this type of approach. This proposed study will evaluate a more intermediate change in practice, primarily geared towards the large number of providers who routinely provide transvaginal ultrasound. For those providers, moving from TVS to TAS could be both cost effective and acceptable to patients.

In detail, the study will enroll patients presenting for medical abortion at multiple clinical sites. These women will undergo routine intake per usual clinical protocol, then randomized to receive either TVS or TAS. Afterwards, routine clinical care will be provided by the clinician, which can include medical abortion provision or further testing to determine eligibility. Women will complete an acceptability survey at the conclusion of the visit.

For providers, prior to participation, providers will complete a questionnaire regarding professional characteristics. Investigators will provide a training session for all providers at each site to review TAS (i.e., techniques and standardized reporting) assuming some providers have less experience with this when compared to TVS in early pregnancy. This training session will help minimize differences in TVS and TAS related to provider experience or variability in current practice. In addition, prior to participant enrollment, each clinic site will enroll 5 pilot patients, during which providers will perform only TAS to accustom providers and clinic staff to study protocols. Each clinician will perform TAS on at least 2 but no more than 5 pilot patients.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish- speaking women seeking medical abortion
* 18 years or older
* Women at an estimated gestational age up to 70 days from last menstrual period (LMP)

Exclusion Criteria:

* Women under 18 years old
* Women at an estimated gestational age greater than 70 days from LMP at enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Westhoff, MD MSc, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Planned Parenthood of Northern, Central, and Southern New Jersey, Morristown, New Jersey
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pazol K, Creanga AA, Burley KD, Jamieson DJ. Abortion surveillance - United States, 2011. MMWR Surveill Summ. 2014 Nov 28;63(11):1-41. PMID 25426741
- [Background] Pazol K, Creanga AA, Zane SB. Trends in use of medical abortion in the United States: reanalysis of surveillance data from the Centers for Disease Control and Prevention, 2001-2008. Contraception. 2012 Dec;86(6):746-51. doi: 10.1016/j.contraception.2012.05.023. Epub 2012 Jul 6. PMID 22770796
- [Background] Jordan B, Shields WC. Happy anniversary mifepristone: a decade of promise and challenges. Contraception. 2010 Sep;82(3):219-20. doi: 10.1016/j.contraception.2010.05.017. No abstract available. PMID 20705148
- [Background] Finer LB, Wei J. Effect of mifepristone on abortion access in the United States. Obstet Gynecol. 2009 Sep;114(3):623-630. doi: 10.1097/AOG.0b013e3181b2a74d. PMID 19701044
- [Background] Raymond EG, Grossman D, Wiebe E, Winikoff B. Reaching women where they are: eliminating the initial in-person medical abortion visit. Contraception. 2015 Sep;92(3):190-3. doi: 10.1016/j.contraception.2015.06.020. Epub 2015 Jun 29. PMID 26134280
- [Background] Chong E, Frye LJ, Castle J, Dean G, Kuehl L, Winikoff B. A prospective, non-randomized study of home use of mifepristone for medical abortion in the U.S. Contraception. 2015 Sep;92(3):215-9. doi: 10.1016/j.contraception.2015.06.026. Epub 2015 Jul 2. PMID 26142620
- [Background] Gold M, Chong E. If we can do it for misoprostol, why not for mifepristone? The case for taking mifepristone out of the office in medical abortion. Contraception. 2015 Sep;92(3):194-6. doi: 10.1016/j.contraception.2015.06.011. Epub 2015 Jun 18. PMID 26093187
- [Background] Grossman D, Goldstone P. Mifepristone by prescription: a dream in the United States but reality in Australia. Contraception. 2015 Sep;92(3):186-9. doi: 10.1016/j.contraception.2015.06.014. Epub 2015 Jun 19. PMID 26096369
- [Background] Harper C, Ellertson C, Winikoff B. Could American women use mifepristone-misoprostol pills safely with less medical supervision? Contraception. 2002 Feb;65(2):133-42. doi: 10.1016/s0010-7824(01)00300-6. PMID 11927116
- [Background] Foster AM, Jackson CB, LaRoche KJ, Simmonds K, Taylor D. From qualified physician to licensed health care professional: the time has come to change mifepristone's label. Contraception. 2015 Sep;92(3):200-2. doi: 10.1016/j.contraception.2015.06.022. Epub 2015 Jun 30. No abstract available. PMID 26134281
- [Background] Kopp Kallner H, Gomperts R, Salomonsson E, Johansson M, Marions L, Gemzell-Danielsson K. The efficacy, safety and acceptability of medical termination of pregnancy provided by standard care by doctors or by nurse-midwives: a randomised controlled equivalence trial. BJOG. 2015 Mar;122(4):510-7. doi: 10.1111/1471-0528.12982. Epub 2014 Jul 18. PMID 25040643
- [Background] Warriner IK, Wang D, Huong NT, Thapa K, Tamang A, Shah I, Baird DT, Meirik O. Can midlevel health-care providers administer early medical abortion as safely and effectively as doctors? A randomised controlled equivalence trial in Nepal. Lancet. 2011 Apr 2;377(9772):1155-61. doi: 10.1016/S0140-6736(10)62229-5. PMID 21458058
- [Background] Bennett IM, Baylson M, Kalkstein K, Gillespie G, Bellamy SL, Fleischman J. Early abortion in family medicine: clinical outcomes. Ann Fam Med. 2009 Nov-Dec;7(6):527-33. doi: 10.1370/afm.1051. PMID 19901312
- [Background] Prine LW, Lesnewski R. Medication abortion and family physicians' scope of practice. J Am Board Fam Pract. 2005 Jul-Aug;18(4):304-6. doi: 10.3122/jabfm.18.4.304. No abstract available. PMID 15994476
- [Background] Prine L, Shannon C, Gillespie G, Crowden WA, Fortin J, Howe M, Dzuba I. Medical abortion: outcomes in a family medicine setting. J Am Board Fam Med. 2010 Jul-Aug;23(4):509-13. doi: 10.3122/jabfm.2010.04.090229. PMID 20616293
- [Background] Wu JP, Godfrey EM, Prine L, Andersen KL, MacNaughton H, Gold M. Women's satisfaction with abortion care in academic family medicine centers. Fam Med. 2015 Feb;47(2):98-106. PMID 25646981
- [Background] Grossman D, Grindlay K. Alternatives to ultrasound for follow-up after medication abortion: a systematic review. Contraception. 2011 Jun;83(6):504-10. doi: 10.1016/j.contraception.2010.08.023. Epub 2010 Oct 8. PMID 21570546
- [Background] Blum J, Shochet T, Lynd K, Lichtenberg ES, Fischer D, Arnesen M, Winikoff B, Blumenthal PD. Can at-home semi-quantitative pregnancy tests serve as a replacement for clinical follow-up of medical abortion? A US study. Contraception. 2012 Dec;86(6):757-62. doi: 10.1016/j.contraception.2012.06.005. Epub 2012 Aug 13. PMID 22895097
- [Background] Bracken H, Lohr PA, Taylor J, Morroni C, Winikoff B. RU OK? The acceptability and feasibility of remote technologies for follow-up after early medical abortion. Contraception. 2014 Jul;90(1):29-35. doi: 10.1016/j.contraception.2014.03.016. Epub 2014 Apr 13. PMID 24815098
- [Background] Michie L, Cameron ST. Simplified follow-up after early medical abortion: 12-month experience of a telephone call and self-performed low-sensitivity urine pregnancy test. Contraception. 2014 May;89(5):440-5. doi: 10.1016/j.contraception.2014.01.010. Epub 2014 Jan 21. PMID 24560481
- [Background] Oppegaard KS, Qvigstad E, Fiala C, Heikinheimo O, Benson L, Gemzell-Danielsson K. Clinical follow-up compared with self-assessment of outcome after medical abortion: a multicentre, non-inferiority, randomised, controlled trial. Lancet. 2015 Feb 21;385(9969):698-704. doi: 10.1016/S0140-6736(14)61054-0. Epub 2014 Oct 30. PMID 25468164
- [Background] Clark WH, Gold M, Grossman D, Winikoff B. Can mifepristone medical abortion be simplified? A review of the evidence and questions for future research. Contraception. 2007 Apr;75(4):245-50. doi: 10.1016/j.contraception.2006.11.011. Epub 2007 Jan 18. PMID 17362700
- [Background] Rogo K. Improving technologies to reduce abortion-related morbidity and mortality. Int J Gynaecol Obstet. 2004 Jun;85 Suppl 1:S73-82. doi: 10.1016/j.ijgo.2004.02.010. PMID 15147856
- [Background] Cleland K, Smith N. Aligning mifepristone regulation with evidence: driving policy change using 15 years of excellent safety data. Contraception. 2015 Sep;92(3):179-81. doi: 10.1016/j.contraception.2015.06.016. Epub 2015 Jun 18. No abstract available. PMID 26093188
- [Background] Wade VA, Karnon J, Elshaug AG, Hiller JE. A systematic review of economic analyses of telehealth services using real time video communication. BMC Health Serv Res. 2010 Aug 10;10:233. doi: 10.1186/1472-6963-10-233. PMID 20696073
- [Background] Gomperts RJ, Jelinska K, Davies S, Gemzell-Danielsson K, Kleiverda G. Using telemedicine for termination of pregnancy with mifepristone and misoprostol in settings where there is no access to safe services. BJOG. 2008 Aug;115(9):1171-5; discussion 1175-8. doi: 10.1111/j.1471-0528.2008.01787.x. Epub 2008 Jul 10. PMID 18637010
- [Background] Gomperts R, van der Vleuten K, Jelinska K, da Costa CV, Gemzell-Danielsson K, Kleiverda G. Provision of medical abortion using telemedicine in Brazil. Contraception. 2014 Feb;89(2):129-33. doi: 10.1016/j.contraception.2013.11.005. Epub 2013 Nov 12. PMID 24314910
- [Background] Wiebe ER. Use of telemedicine for providing medical abortion. Int J Gynaecol Obstet. 2014 Feb;124(2):177-8. doi: 10.1016/j.ijgo.2013.07.038. Epub 2013 Nov 15. No abstract available. PMID 24332519
- [Background] Grossman DA, Grindlay K, Buchacker T, Potter JE, Schmertmann CP. Changes in service delivery patterns after introduction of telemedicine provision of medical abortion in Iowa. Am J Public Health. 2013 Jan;103(1):73-8. doi: 10.2105/AJPH.2012.301097. Epub 2012 Nov 15. PMID 23153158
- [Background] Grossman D, Grindlay K, Buchacker T, Lane K, Blanchard K. Effectiveness and acceptability of medical abortion provided through telemedicine. Obstet Gynecol. 2011 Aug;118(2 Pt 1):296-303. doi: 10.1097/AOG.0b013e318224d110. PMID 21775845
- [Background] Grindlay K, Lane K, Grossman D. Women's and providers' experiences with medical abortion provided through telemedicine: a qualitative study. Womens Health Issues. 2013 Mar-Apr;23(2):e117-22. doi: 10.1016/j.whi.2012.12.002. Epub 2013 Feb 12. PMID 23410620
- [Background] Atrash HK, MacKay HT, Hogue CJ. Ectopic pregnancy concurrent with induced abortion: incidence and mortality. Am J Obstet Gynecol. 1990 Mar;162(3):726-30. doi: 10.1016/0002-9378(90)90995-j. PMID 2316578
- [Background] Shannon C, Brothers LP, Philip NM, Winikoff B. Ectopic pregnancy and medical abortion. Obstet Gynecol. 2004 Jul;104(1):161-7. doi: 10.1097/01.AOG.0000130839.61098.12. PMID 15229016
- [Background] Cleland K, Creinin MD, Nucatola D, Nshom M, Trussell J. Significant adverse events and outcomes after medical abortion. Obstet Gynecol. 2013 Jan;121(1):166-71. doi: 10.1097/aog.0b013e3182755763. PMID 23262942
- [Background] Practice bulletin no. 143: medical management of first-trimester abortion. Obstet Gynecol. 2014 Mar;123(3):676-692. doi: 10.1097/01.AOG.0000444454.67279.7d. PMID 24553166
- [Background] Kapp N, Whyte P, Tang J, Jackson E, Brahmi D. A review of evidence for safe abortion care. Contraception. 2013 Sep;88(3):350-63. doi: 10.1016/j.contraception.2012.10.027. Epub 2012 Dec 20. PMID 23261233
- [Background] Elul B, Hajri S, Ngoc NN, Ellertson C, Slama CB, Pearlman E, Winikoff B. Can women in less-developed countries use a simplified medical abortion regimen? Lancet. 2001 May 5;357(9266):1402-5. doi: 10.1016/s0140-6736(00)04563-3. PMID 11356438
- [Background] Coyaji K, Elul B, Krishna U, Otiv S, Ambardekar S, Bopardikar A, Raote V, Ellertson C, Winikoff B. Mifepristone-misoprostol abortion: a trial in rural and urban Maharashtra, India. Contraception. 2002 Jul;66(1):33-40. doi: 10.1016/s0010-7824(02)00309-8. PMID 12169379
- [Background] Mundle S, Elul B, Anand A, Kalyanwala S, Ughade S. Increasing access to safe abortion services in rural India: experiences with medical abortion in a primary health center. Contraception. 2007 Jul;76(1):66-70. doi: 10.1016/j.contraception.2007.03.010. Epub 2007 May 25. PMID 17586140
- [Background] Louie KS, Tsereteli T, Chong E, Aliyeva F, Rzayeva G, Winikoff B. Acceptability and feasibility of mifepristone medical abortion in the early first trimester in Azerbaijan. Eur J Contracept Reprod Health Care. 2014 Dec;19(6):457-64. doi: 10.3109/13625187.2014.933956. Epub 2014 Jul 22. PMID 25047120
- [Background] Louie KS, Chong E, Tsereteli T, Avagyan G, Vardanyan S, Winikoff B. The introduction of first trimester medical abortion in Armenia. Reprod Health Matters. 2015 Feb;22(44 Suppl 1):56-66. doi: 10.1016/S0968-8080(15)43824-8. PMID 25702069
- [Background] Ellertson C, Elul B, Ambardekar S, Wood L, Carroll J, Coyaji K. Accuracy of assessment of pregnancy duration by women seeking early abortions. Lancet. 2000 Mar 11;355(9207):877-81. doi: 10.1016/S0140-6736(99)10170-3. PMID 10752703
- [Background] Savitz DA, Terry JW Jr, Dole N, Thorp JM Jr, Siega-Riz AM, Herring AH. Comparison of pregnancy dating by last menstrual period, ultrasound scanning, and their combination. Am J Obstet Gynecol. 2002 Dec;187(6):1660-6. doi: 10.1067/mob.2002.127601. PMID 12501080
- [Background] McGalliard C, Gaudoin M. Routine ultrasound for pregnancy termination requests increases women's choice and reduces inappropriate treatments. BJOG. 2004 Jan;111(1):79-82. doi: 10.1111/j.1471-0528.2004.00014.x. PMID 14687056
- [Background] Blanchard K, Cooper D, Dickson K, Cullingworth L, Mavimbela N, von Mollendorf C, van Bogaert LJ, Winikoff B. A comparison of women's, providers' and ultrasound assessments of pregnancy duration among termination of pregnancy clients in South Africa. BJOG. 2007 May;114(5):569-75. doi: 10.1111/j.1471-0528.2007.01293.x. PMID 17439565
- [Background] Bracken H, Clark W, Lichtenberg ES, Schweikert SM, Tanenhaus J, Barajas A, Alpert L, Winikoff B. Alternatives to routine ultrasound for eligibility assessment prior to early termination of pregnancy with mifepristone-misoprostol. BJOG. 2011 Jan;118(1):17-23. doi: 10.1111/j.1471-0528.2010.02753.x. Epub 2010 Nov 23. PMID 21091926
- [Background] Raymond EG, Bracken H. Early medical abortion without prior ultrasound. Contraception. 2015 Sep;92(3):212-4. doi: 10.1016/j.contraception.2015.04.008. Epub 2015 Apr 24. PMID 25916975
- [Background] Fielding SL, Schaff EA, Nam NY. Clinicians' perception of sonogram indication for mifepristone abortion up to 63 days. Contraception. 2002 Jul;66(1):27-31. doi: 10.1016/s0010-7824(02)00316-5. PMID 12169378
- [Background] Schonberg D, Wang LF, Bennett AH, Gold M, Jackson E. The accuracy of using last menstrual period to determine gestational age for first trimester medication abortion: a systematic review. Contraception. 2014 Nov;90(5):480-7. doi: 10.1016/j.contraception.2014.07.004. Epub 2014 Jul 18. PMID 25152258
- [Background] Kaneshiro B, Edelman A, Sneeringer RK, Ponce de Leon RG. Expanding medical abortion: can medical abortion be effectively provided without the routine use of ultrasound? Contraception. 2011 Mar;83(3):194-201. doi: 10.1016/j.contraception.2010.07.023. Epub 2010 Sep 17. PMID 21310279
- [Background] Kulier R, Kapp N. Comprehensive analysis of the use of pre-procedure ultrasound for first- and second-trimester abortion. Contraception. 2011 Jan;83(1):30-3. doi: 10.1016/j.contraception.2010.06.014. Epub 2010 Aug 5. PMID 21134500
- [Background] Lohr PA, Reeves MF, Creinin MD. A comparison of transabdominal and transvaginal ultrasonography for determination of gestational age and clinical outcomes in women undergoing early medical abortion. Contraception. 2010 Mar;81(3):240-4. doi: 10.1016/j.contraception.2009.10.008. Epub 2009 Nov 14. PMID 20159181
- [Background] Braithwaite JM, Economides DL. Acceptability by patients of transvaginal sonography in the elective assessment of the first-trimester fetus. Ultrasound Obstet Gynecol. 1997 Feb;9(2):91-3. doi: 10.1046/j.1469-0705.1997.09020091.x. PMID 9132262
- [Background] Rosati P, Guariglia L. Acceptability of early transvaginal or abdominal sonography in the first half of pregnancy. Arch Gynecol Obstet. 2000 Sep;264(2):80-3. doi: 10.1007/s004040000085. PMID 11045328
- [Background] Dutta RL, Economides DL. Patient acceptance of transvaginal sonography in the early pregnancy unit setting. Ultrasound Obstet Gynecol. 2003 Nov;22(5):503-7. doi: 10.1002/uog.892. PMID 14618664
- [Result] Fu A, Weber CE, Gilmore E, Davis AR, Hirsch G, Westhoff CL. A noninferiority randomized controlled trial to compare transabdominal and transvaginal sonography for eligibility assessment prior to medical abortion. Contraception. 2018 Sep;98(3):199-204. doi: 10.1016/j.contraception.2018.05.005. Epub 2018 May 9. PMID 29752922

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were excluded from the analysis due to study withdrawal prior to receiving sonography.
Groups:
- Transabdominal Sonography: Subjects will receive transabdominal sonography using a standard ultrasound device to determine medical abortion eligibility.
  A transabdominal ultrasound is used to look at the pelvic organs. Gel is placed on your abdomen. Then a small, handheld unit called a transducer is gently moved around to view the pelvic organs. The transducer sound waves make a picture on the TV screen.
  Transabdominal sonography: Ultrasound machines vary by site. At Planned Parenthood and Columbia University Medical Center, providers utilize the LOGIQ P5 ultrasound machine, manufactured by General Electric Healthcare.
- Transvaginal Sonography: Subjects will receive transvaginal sonography using a standard ultrasound device to determine medical abortion eligibility.
  Transvaginal ultrasound is an examination of the female pelvis and urogenital tract (kidneys and bladder). It differs from an abdominal ultrasound as it looks at the pelvic organs from inside the vagina.
  Transvaginal sonography: Ultrasound machines vary by site. At Planned Parenthood and Columbia University Medical Center, providers utilize the LOGIQ P5 ultrasound machine, manufactured by General Electric Healthcare.
Period: Overall Study
Arm/Group | Transabdominal Sonography | Transvaginal Sonography
Started | 319 | 315
Completed | 317 | 312
Not Completed | 2 | 3
Not completed — Did not receive TAS | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Probe malfunction | 0 | 1
Not completed — Ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transabdominal Sonography | Transvaginal Sonography | Total
Number analyzed (Participants) | 317 | 312 | 629
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 317 | 312 | 629
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 317 | 312 | 629
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 179 | 168 | 347
  Not Hispanic or Latino | 114 | 123 | 237
  Unknown or Not Reported | 24 | 21 | 45
Region of Enrollment [Number; unit: participants]
  United States | 317 | 312 | 629
BMI category [Count of Participants; unit: Participants]
  <25 kg/m^2 | 143 | 135 | 278
  25 - <30 kg/m^2 | 99 | 82 | 181
  30 - <35 kg/m^2 | 49 | 51 | 100
  >35 kg/m^2 | 17 | 38 | 55
  Missing | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects in Each Ultrasound Group With Additional Testing
Description: Evaluate how often a provider orders additional testing prior to medical abortion, but after either 1) patient history and TAS or 2) patient history and TVS.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Transabdominal Sonography | Transvaginal Sonography
Number analyzed (Participants) | 317 | 312
Participants | 63 | 14

2. Primary Outcome: Visual Analog Scale (VAS) Score for Patient Acceptability for Either Modality of Ultrasound
Description: To measure patient satisfaction after ultrasound examination, each participant will complete an acceptability questionnaire regarding the type of ultrasound she received (TVS or TAS) using a visual analog scale (VAS). The score is on a scale range of 0-100, with 0 being "unacceptable" and 100 being "acceptable." Thus, higher scores are better.
Time Frame: 1 day
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Transabdominal Sonography | Transvaginal Sonography
Number analyzed (Participants) | 317 | 312
score on a scale | 95.9 [17 to 100] | 90.0 [0 to 100]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Transabdominal Sonography | Transvaginal Sonography
All-Cause Mortality (participants affected / at risk) | 0/317 | 0/312
Serious Adverse Events (participants affected / at risk) | 0/317 | 0/312
Other Adverse Events (participants affected / at risk) | 0/317 | 0/312

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT03047551/Prot_SAP_000.pdf